CLINICAL TRIAL: NCT06402071
Title: Clinical Value of the Developed Scoring Systems for Predicting Spontaneous Bacterial Peritonitis in Cirrhotic Ascites
Status: Recruiting | Type: Observational
Sponsor: Dalia Nasser Mohamed (Other)
Responsible Party: Sponsor-Investigator, Dalia Nasser Mohamed, Resident doctor at tropical medicine and gastroenterology department sohag university hospitals, Sohag University
Organization: Sohag University (Other)
Other Study IDs: Soh-Med-24-03-05MS
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Cirrhotic Ascitic Patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A (Cases): Cirrhotic ascitic patients with spontaneous bacterial peritonitis
  Interventions: Diagnostic Test: Ascitic fluid study
- Group B (Controls): Cirrhotic ascitic patients without spontaneous bacterial peritonitis
  Interventions: Diagnostic Test: Ascitic fluid study

INTERVENTIONS:
Diagnostic Test: Ascitic fluid study — Ascitic fluid study will be obtained from all participants
  Other Names: Abdominal ultrasound, liver functions

SUMMARY:
Liver cirrhosis is the clinical end stage of different entities of chronic liver disease when patients suffer from considerable mortality and morbidity, both of which are correlated positively with disease severity. Ascites are the most common complication, and around 60% of patients with compensated cirrhosis develop ascites within 10 years of disease onset (D'Amico et al., 2015).

Spontaneous bacterial peritonitis (SBP) which is defined by acute infection of ascitic fluid, an abnormal accumulation of fluid in the abdomen without a distinct or identifiable source of infection, with ascitic fluid absolute neutrophil count >250 cells/mm³, whether or not there is culture growth. is a major cause of morbidity and mortality in cirrhotic patients with ascites. SBP is estimated to affect 10-30% of cirrhotic patients hospitalized with ascites, and mortality in this group approaches 30%. Many of these patients are asymptomatic, and it is therefore recommended that all patients with ascites undergo paracentesis at the time of admission to confirm the SBP status. Although SBP is less prevalent in an outpatient setting, it is reasonable to also evaluate the ascitic fluid of outpatients because of the high mortality associated with SBP Platelets are considered an important source of pro-thrombotic agents associated with inflammatory markers and play a role in the initiation and propagation of inflammatory diseases. Platelets with large sizes have many granules that can exert their hemostatic and proinflammatory actions with greater efficiency. For these reasons, the mean platelet volume (MPV) and platelet distribution width (PDW) may be considered indicators of platelet function and activation (Abdelmoez et al., 2016).

MPV and PDW are routine tests that are a part of a complete blood count. An increase in MPV has been observed in chronic viral hepatitis because of an increase in the entry of newly produced platelets into circulation, which are larger in volume than the old platelets (Castellote et al., 2008; Suvak et al., 2013). Therefore, mean platelet volume and platelet distribution width measurement may be used in predicting spontaneous bacterial peritonitis (Gálvez-Martínez et al., 2015; Abdelmoez et al., 2017).

The blood neutrophil-lymphocyte ratio (NLR) is a crucial parameter for the balance of the inflammatory and immune systems, reflecting responses to systemic inflammation In patients with decompensated liver cirrhosis, NLR is a non-invasive marker that can be used to predict the occurrence of hospital infection (Cai et al., 2017), NLR is a predictor of SBP that can be utilized in combination with other markers. According to (Mousa et al., 2016), blood NLR > 2.89 had an 80.3% sensitivity and 88.9% specificity for diagnosing SBP, while blood NLR and CRP combined (cut-off 11.3 mg/dL) had a 95.1% sensitivity and 96.3% specificity (Mousa et al., 2016).

Although single tests have shown some value in predicting SBP, their studies have been small and inconsistent. In order to predict SBP in patients with cirrhotic ascites, prediction scores in conjunction with clinical and laboratory indicators are therefore being developed recently (Dahiya et al., 2023; Wehmeyer et al., 2014).

In summary, Infections are common in liver cirrhosis patients, and SBP is one of the most prevalent, with varying frequency but a significant fatality rate. One of the most crucial factors in treating this significant consequence of decompensated liver cirrhosis is early detection. Finding non-invasive, affordable, and simple-to-implement parameters related to SBP that have a predictive role is essential. However, need to be kept in mind these methods cannot completely replace paracentesis, more studies are needed to determine whether non-invasive methods are sufficiently accurate to identify the development of SBP in cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* All cirrhotic patients with ascites with or without spontaneous bacterial peritonitis, SBP that is defined as ascites PMN count >250 cells /mm3, without evidence of inta-abdominal surgical cause of infection) will be included in the study.

Exclusion Criteria:

* Patients with ascites because of causes other than cirrhosis, such as renal, cardiac, nutritional, tuberculosis, peritoneal carcinomatosis.

If there is evidence of intra or extrahepatic malignancy. If there is evidence of other non-infectious inflammatory conditions like rheumatoid arthritis, ankylosing spondylitis and /or auto immune diseases.

If there are infections other than SBP, such as pneumonia, urinary tract infection, and skin infection.

Patients receiving anticoagulants, oral contraception or NSAIDs before hospital admission.

Patients on recent usage of antibiotics prior to hospital admission. If there is evidence of monomicrobial non-neutrocytic bacterascites when PMNL count is <250/mm3 and the culture positive while the patient may present with symptoms and signs of infection.

Patients with secondary peritonitis which is described as the presence of a very high PMNL count with a lack of response to antibiotic treatment or glucose level in ascitic fluid <50 mg/dl, protein >10 g/l or suspected intraabdominal surgical cause of infection.

Patients with diseases associated with increased MPV, for example, diabetes mellitus, cardiovascular disease, hyperthyroidism, immune thrombocytopenia, and myeloproliferative disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This case control study will include Patients with liver cirrhosis diagnosed by combination of clinical, sonographic and laboratory data admitted to Sohag University hospital with ascites with or without evidence of ascitic fluid infection.
  According to the ascitic fluid analysis patients will be divided according to the polymorphnuclear cells count in the ascitic fluid into two groups:
  1. Group I: will include cirrhotic ascitic patients with SBP.
  2. Group II: will include age matched ci
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
-Determine the cases of SBP among all cirrhotic patients with ascites | 1 year
  compare role of markers of systemic inflammatory response individually or built in model scores as non- invasive predictors for SBP

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Galvez-Martinez M, Servin-Caamano AI, Perez-Torres E, Salas-Gordillo F, Rivera-Gutierrez X, Higuera-de la Tijera F. Mean platelet volume as a novel predictor of systemic inflammatory response in cirrhotic patients with culture-negative neutrocytic ascites. World J Hepatol. 2015 May 8;7(7):1001-6. doi: 10.4254/wjh.v7.i7.1001. PMID 25954482
- [Background] Wehmeyer MH, Krohm S, Kastein F, Lohse AW, Luth S. Prediction of spontaneous bacterial peritonitis in cirrhotic ascites by a simple scoring system. Scand J Gastroenterol. 2014 May;49(5):595-603. doi: 10.3109/00365521.2013.848471. Epub 2014 Mar 27. PMID 24673156
- [Background] Abdel-Razik A, Mousa N, Besheer TA, Eissa M, Elhelaly R, Arafa M, El-Wakeel N, Eldars W. Neutrophil to lymphocyte ratio as a reliable marker to predict insulin resistance and fibrosis stage in chronic hepatitis C virus infection. Acta Gastroenterol Belg. 2015 Dec;78(4):386-92. PMID 26712048
- [Background] Metwally K, Fouad T, Assem M, Abdelsameea E, Yousery M. Predictors of Spontaneous Bacterial Peritonitis in Patients with Cirrhotic Ascites. J Clin Transl Hepatol. 2018 Dec 28;6(4):372-376. doi: 10.14218/JCTH.2018.00001. Epub 2018 Jul 18. PMID 30637213